CLINICAL TRIAL: NCT05769842
Title: Can Propofol Reduce Respiratory Adverse Events During Extubation in Children With Tonsillectomy? A Prospective Randomized Controlled Study
Brief Title: Effects of Propofol on Respiratory Adverse Events During Extubation in Children Undergoing Tonsil Adenoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2022-01
Record Dates: First submitted 2023-02-02; First posted 2023-03-15 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Airway Complication of Anesthesia
Keywords: propofol; tracheal extubation; respiratory adverse events
MeSH Terms: interventions — Propofol; Saline Solution

STUDY DESIGN:
Intervention Model Description: Pediatric patients were randomly assigned to either the propofol group or the control group. In the propofol group, after the child regained spontaneous breathing before extubation, propofol was administered in small repeated doses, each dose being 0.5mg/kg, with a total amount of 1~2mg/kg. The control group received an equivalent volume of normal saline. The occurrence of respiratory adverse events (such as laryngospasm, bronchospasm, breath-holding, coughing, decreased oxygen saturation, and airway obstruction) was observed in both groups post-extubation, with the presence of any one or more events considered indicative of respiratory adverse events.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- propofol group (Experimental): Children aged 3 to 8 years who had had their tonsil adenoidectomy were collected. Propofol 3mg/kg, remifentanil 3-5ug /kg and atropine 0.01mg/kg were used for intravenous induction intubation. Sevoflurane was used for intraoperative anesthesia, propartamol 30mg/kg and hydromorphone 5-10ug /kg were used for postoperative analgesia.When sevoflurane was shut down at the end of the operation, oxygen flow was increased to more than 7L/min, and extubation was prepared for spontaneous respiration recovery, propofol was given a small amount of 1~2mg/kg multiple times without inhibition of spontaneous respiration.
  Interventions: Drug: propofol
- control group (Sham Comparator): Anesthesia induction is the same as before.At the end of the operation, sevoflurane was shut down and oxygen flow was increased to more than 7L/min. No other treatment was performed during extubation.
  Interventions: Drug: normal saline

INTERVENTIONS:
Drug: propofol — Propofol was mainly used in the intervention group during anesthesia extubation. Propofol was given a small amount of times about 1~2mg/kg before extubation when the patient recovered spontaneously.
  Other Names: No Other Intervention Names
  Arms: propofol group
Drug: normal saline — Same dose as propofol.
  Other Names: No Other Intervention Names
  Arms: control group

SUMMARY:
The main objective of this study was to investigate whether propofol assisted extubation could reduce the incidence of respiratory adverse events in children with tonsil adenoidectomy.

DETAILED DESCRIPTION:
In pediatric surgery, the incidence of perioperative respiratory adverse events in children undergoing tonsillectomy is higher than that of general surgery. Studies have shown that intravenous induction can reduce perioperative respiratory adverse events compared with inhalation induction. There are also literatures that show that intravenous anesthesia can significantly reduce cough and hemodynamic reactions during the wake period compared with balanced anesthesia.However, inhalation anesthesia is easier to use and can monitor the depth of anesthesia, so it is used more frequently than intravenous anesthesia.The incidence of respiratory adverse events has not been compared between intraoperative sevoflurane maintenance and extubation with a small amount of propofol versus total sevoflurane maintenance and extubation.The objective of this study was to investigate whether propofol can reduce perioperative adverse respiratory events in children undergoing tonsillectomy.

ELIGIBILITY:
Inclusion Criteria:

* age: 3~8 years old,
* general anesthesia for tracheal intubation in ASA Grade I to III patients undergoing tonsil adenoidectomy,
* the operation time is 10~60 minutes,
* sign informed consent.

Exclusion Criteria:

* patients with congenital heart disease, tumor, severe lung disease, liver and kidney function disease, nervous system disease, coagulation dysfunction, etc,
* children who do not consent to the test.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 239 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
respiratory adverse events | From the moment of extubation to the time before entering the resuscitation room, the maximum time is no more than four hours.
  These include six items in total:
  1. laryngeal spasm: little or no airflow in jaw support,need mask pressure ventilation or anesthetic relief .
  2. bronchospasm:airway pressure increased, tidal volume decreased, and lung auscultation and wheezing were observed, accompanied by decreased oxygen saturation.
  3. breath-holding:no breathing time > 5 seconds or more.
  4. cough:0 = no cough; 1 point = weak cough; 2 points = strong cough; 3 points = continuous strong cough.
  5. low oxygen saturation:less than 92% on oxygen.
  6. respiratory obstruction:jaw support is needed for relief.

SECONDARY OUTCOMES:
extubation time | No more than three hours from the end of the procedure until the tracheal tube was pulled out.
  longer than 15 minutes means longer extubation time.
Richmond Agitation Sedation Scale | From the moment of extubation to the time before entering the resuscitation room, the maximum time is no more than four hours.
  The score ranges from -5 to +4. A higher score indicates more agitation and a lower score indicates greater calmness. In this study, a score greater than or equal to 1 indicates agitation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhijian Zhou, Study Director — Children's Hospital of Fudan University
Locations (1):
- Children's Hospital affiliated with Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramgolam A, Hall GL, Zhang G, Hegarty M, von Ungern-Sternberg BS. Inhalational versus IV induction of anesthesia in children with a high risk of perioperative respiratory adverse events. Anesthesiology. 2018;128(6):1065-1074. AORN J. 2018 Nov;108(5):566-571. doi: 10.1002/aorn.12390. No abstract available. PMID 30376178
- [Background] Hohlrieder M, Tiefenthaler W, Klaus H, Gabl M, Kavakebi P, Keller C, Benzer A. Effect of total intravenous anaesthesia and balanced anaesthesia on the frequency of coughing during emergence from the anaesthesia. Br J Anaesth. 2007 Oct;99(4):587-91. doi: 10.1093/bja/aem203. Epub 2007 Jul 27. PMID 17660457
- [Background] von Ungern-Sternberg BS, Davies K, Hegarty M, Erb TO, Habre W. The effect of deep vs. awake extubation on respiratory complications in high-risk children undergoing adenotonsillectomy: a randomised controlled trial. Eur J Anaesthesiol. 2013 Sep;30(9):529-36. doi: 10.1097/EJA.0b013e32835df608. PMID 23344124
- [Derived] Liao R, Zhou Z, Wang X, Shao H. Impact of Propofol Administered before Extubation on Respiratory Adverse Events in Pediatric Patients Undergoing Tonsillectomy and Adenoidectomy: A Randomized Controlled Trial. Br J Hosp Med (Lond). 2024 Nov 30;85(11):1-15. doi: 10.12968/hmed.2024.0431. Epub 2024 Nov 18. PMID 39618204